CLINICAL TRIAL: NCT01652092
Title: Allogeneic Hematopoietic Stem Cell Transplant for Patients With Primary Immune Deficiencies
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012OC055; MT2012-10C (Other: Blood and Marrow Transplantation Program)
Record Dates: First submitted 2012-07-25; First posted 2012-07-27 (Estimated); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: SCID; Omenn's Syndrome; Reticular Dysgenesis; Wiskott-Aldrich Syndrome; Bare Lymphocyte Syndrome; Common Variable Immunodeficiency; Chronic Granulomatous Disease; CD40 Ligand Deficiency; Hyper IgM Syndrome; X-linked Lymphoproliferative Disease; Hemophagocytic Lymphohistiocytosis; Griscelli Syndrome; Chediak-Higashi Syndrome; Langerhan's Cell Histiocytosis
Keywords: immunodeficiency disorder; histiocytic disorder
MeSH Terms: conditions — Severe Combined Immunodeficiency; Reticular dysgenesis; Wiskott-Aldrich Syndrome; Common Variable Immunodeficiency; Granulomatous Disease, Chronic; Hyper-IgM Immunodeficiency Syndrome; Lymphoproliferative Disorders; Lymphohistiocytosis, Hemophagocytic; Chediak-Higashi Syndrome; Histiocytosis, Langerhans-Cell; Immunologic Deficiency Syndromes | interventions — Alemtuzumab; Cyclophosphamide; Busulfan; Stem Cell Transplantation; fludarabine phosphate; Melphalan; Mesna; Sodium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Arm A: Fully Myeloablative regimen (Other): For use in patients with diseases including Wiskott-Aldrich syndrome, MHC Class II deficiency, hypomorphic SCID, etc. Receives Alemtuzumab 0.3 mg/kg intravenously (IV) on days -12 through -10, cyclophosphamide 50 mg/kg IV plus MESNA on days -9 through -6, busulfan 0.8 or 1.1 mg/kg IV on days -5 through -2 and stem cell infusion on day 0.
  Interventions: Drug: Alemtuzumab 0.3 mg; Drug: Cyclophosphamide; Drug: Busulfan; Biological: Stem Cell Transplantation; Drug: MESNA
- Arm B: Reduced Toxicity Ablative Regimen (Other): For use in patients with diseases including SCID, CGD, CHS and other CID. Receives Alemtuzumab 0.3 mg/kg intravenously (IV) on days -12 through -10, busulfan 0.8 or 1.1 mg/kg IV on days -9 through -6, fludarabine phosphate 40 mg/m^2 IV on days -5 through -2 and stem cell infusion on day 0.
  Interventions: Drug: Alemtuzumab 0.3 mg; Biological: Stem Cell Transplantation; Drug: Fludarabine phosphate 40 mg; Drug: Busulfan
- Arm C: Reduced Intensity Conditioning (Other): For use in patients with diseases including HLH. Receives Alemtuzumab 0.2 mg/kg intravenously (IV) on days -14 through -10, fludarabine phosphate 30 mg/m^2 IV on days -8 through -4, melphalan 140 mg/m^2 IV on day -3 and stem cell infusion on day 0.
  Interventions: Biological: Stem Cell Transplantation; Drug: Melphalan; Drug: Alemtuzumab 0.2 mg; Drug: Fludarabine phosphate 30 mg
- Arm D: No Preparative Regimen (Other): For use in patients with complete SCID phenotype with no evidence of maternal engraftment or residual immune function who will be receiving their stem cell transplantation from a genotypically matched donor.
  Interventions: Biological: Stem Cell Transplantation

INTERVENTIONS:
Drug: Alemtuzumab 0.3 mg — 0.3 mg/kg intravenously (IV) on days -12 through -10
  Other Names: Campath-1H
  Arms: Arm A: Fully Myeloablative regimen; Arm B: Reduced Toxicity Ablative Regimen
Drug: Cyclophosphamide — cyclophosphamide 50 mg/kg IV on days -9 through -6
  Other Names: Cytoxan
  Arms: Arm A: Fully Myeloablative regimen
Drug: Busulfan — busulfan 0.8 or 1.1 mg/kg IV on days -5 through -2
  Other Names: Myerlan
  Arms: Arm A: Fully Myeloablative regimen
Biological: Stem Cell Transplantation — Unrelated donor bone marrow will be collected in the usual manner using established parameters determined by the National Marrow Donor Program. A minimum of 3 x 10^8 nucleated cells/kg recipient weight will be collected with a goal of ≥ 5 x 10^8 nucleated cells/kg recipient weight.
  Umbilical cord blood selection will be per the current University of Minnesota Cord Blood Unit Selection algorithm. One or two units may be used to obtain the minimum cell dose. One of the UCB units selected for transplantation must contain ≥ 3.5 x 10^7 nucleated cells/kg recipient weight based on cell numbers at time of cryopreservation, and the total combined cell dose of both units must be > 5.0 x 10^7 nucleated cells/kg.
Drug: Fludarabine phosphate 40 mg — 40 mg/m^2 IV on days -5 through -2 (for children < 6 months and/or < 10 kg weight dose at 1.33 mg/kg)
  Other Names: Fludara
  Arms: Arm B: Reduced Toxicity Ablative Regimen
Drug: Melphalan — 140 mg/m^2 IV on day -3
  Other Names: Alkeran
  Arms: Arm C: Reduced Intensity Conditioning
Drug: Alemtuzumab 0.2 mg — 0.2 mg/kg intravenously (IV) on days -14 through -10
  Other Names: Campath 1-H
  Arms: Arm C: Reduced Intensity Conditioning
Drug: Busulfan — busulfan 0.8 or 1.1 mg/kg IV on days -9 through -6
  Other Names: Myerlan
  Arms: Arm B: Reduced Toxicity Ablative Regimen
Drug: Fludarabine phosphate 30 mg — fludarabine 30 mg/m^2 IV on days -8 through -4
  Other Names: Fludara
  Arms: Arm C: Reduced Intensity Conditioning
Drug: MESNA — administered as per the standard institutional protocol.
  Other Names: mercaptoethane sulfonate Na (Na being the symbol for sodium); Mesnex
  Arms: Arm A: Fully Myeloablative regimen

SUMMARY:
This is a standard of care treatment guideline for allogeneic hematopoetic stem cell transplant (HSCT) in patients with primary immune deficiencies.

DETAILED DESCRIPTION:
Based on diagnosis and clinical history, a determination of the most appropriate regimen will be made based on the following prep plans:

Arm A: Fully Myeloablative Preparative Regimen, Arm B: Reduced Toxicity Ablative Preparative Regimen, Arm C: Reduced Intensity Conditioning, Arm D: No Preparative Regimen

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of immunodeficiency or histiocytic disorder including the following:

  * Severe combined immunodeficiency (SCID - all variants)
  * Second bone marrow transplant (BMT) for SCID (after graft rejection)
  * Omenn's Syndrome
  * Reticular dysgenesis
  * Wiskott-Aldrich syndrome
  * Major histocompatibility complex (MHC) Class II deficiency (bare lymphocyte syndrome)
  * Hyper IgM Syndrome (CD40 Ligand Deficiency)
  * Common variable immunodeficiency (CVID) with severe phenotype
  * Chronic Granulomatous Disease (CGD)
  * Other severe Combined Immune Deficiencies (CID)
  * Hemophagocytic Lymphohistiocytosis (HLH)
  * X-linked Lymphoproliferative Disease (XLP)
  * Chediak-Higashi Syndrome (CHS)
  * Griscelli Syndrome
  * Langerhans Cell Histiocytosis (LCH)
* Acceptable stem cell sources include:

  * HLA identical or 1 antigen matched sibling donor eligible to donate bone marrow
  * HLA identical or up to a 1 antigen mismatched unrelated BM donor
  * Sibling donor cord blood with acceptable HLA match and cell dose as per current institutional standards
  * Single unrelated umbilical cord blood unit with 0-2 antigen mismatch and minimum cell dose of >5 x 10^7 nucleated cells/kg as per current institutional guidelines
  * Double unrelated umbilical cord blood units that are:

    * up to 2 antigen mismatched to the patient
    * up to 2 antigen mismatched to each other
    * minimum cell dose of at least one single unit must be ≥ 3.5 x 10^7 nucleated cells/kg
    * combined dose of both units must provide a total cell dose of ≥ 5 x 10^7 nucleated cells/kg
* Age: 0 to 50 years
* Adequate organ function and performance status.

Exclusion Criteria

* pregnant or breastfeeding
* active, uncontrolled infection and/or HIV positive
* acute hepatitis or evidence of moderate or severe portal fibrosis or cirrhosis on biopsy

Max Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 57 (Actual)
Dates: Start 2012-09-04 (Actual); Primary Completion 2025-12-30 (Actual); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Neutrophil Engraftment | Day 42
  Neutrophil engraftment is defined as the first day of three consecutive days where the neutrophil count (absolute neutrophil count) is 500 cells/mm3 (0.5 x 109/L) or greater.

SECONDARY OUTCOMES:
Incidence of Graft Failure | Day 100
  Graft failure is defined as not accepting donated cells. The donated cells do not make the new white blood cells, red blood cells and platelets.
Incidence of Chimerism | Day 100, 6 Months, 1 Year
  a state in bone marrow transplantation in which bone marrow and host cells exist compatibly without signs of graft-versus-host rejection disease.
Incidence of Acute Graft-Versus-Host Disease | Day 100
  Acute Graft-Versus-Host Disease is a severe short-term complication created by infusion of donor cells into a foreign host.
Incidence of Chronic Graft-Versus-Host Disease | 6 Months and 1 Year
  Chronic Graft-Versus-Host Disease is a severe long-term complication created by infusion of donor cells into a foreign host.
Incidence of Transplant-Related Mortality | 6 Months
  In the field of transplantation, toxicity is high and all deaths without previous relapse or progression are usually considered as related to transplantation.
Disease-Free Survival | 6 Months
  the length of time after treatment ends that a patient survives without any signs or symptoms of that cancer or any other type of cancer. In a clinical trial, measuring the disease-free survival is one way to see how well a new treatment works.
Overall Survival | 6 Months
  Overall survival will be defined as time from enrollment to date of death or censored at the date of last documented contact for patients still alive.

CONTACTS AND LOCATIONS:
Overall Officials: Christen Ebens, MD, Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (1):
- Masonic Cancer Center, University of Minnesota, Minneapolis, Minnesota, United States